CLINICAL TRIAL: NCT04143191
Title: Sorafenib Plus Transarterial Chemoembolization Versus Sorafenib Alone as Postoperative Adjuvant Treatment for Resectable Primary Advanced Hepatocellular Carcinoma: A Phase 3, Multicenter, Randomized Controlled Trial
Brief Title: Sorafenib Plus TACE Versus Sorafenib Alone as Postoperative Adjuvant Treatment for Resectable Primary Advanced HCC
Acronym: SOURCE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Vice-president, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FAH-20190358
Record Dates: First submitted 2019-10-26; First posted 2019-10-29 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sorafenib (Active Comparator): Patients in this arm will take Sorafenib orally with the dose of 400mg bid on the third day after randomization till recurrence or the end of this trial. If any drug related adverse event occurred, the dosage will be reduced.
  Interventions: Drug: Sorafenib
- Sorafenib plus TACE (Experimental): Patients in this arm will take Sorafenib orally with the dose of 400mg bid on the third day after randomization till recurrence or the end of this trial. TACE will be performed on the fourth day after randomization. If any drug related adverse event occurred, the dosage will be reduced.
  Interventions: Drug: Sorafenib; Procedure: Transarterial chemoembolization

INTERVENTIONS:
Drug: Sorafenib — Sorafenib is one of tyrosine kinase inhibitors. The initial dosage is 400mg orally, twice daily.
Procedure: Transarterial chemoembolization — TACE including conventional TACE (cTACE) and DEB-TACE. Treatment choices are according to the specific condition of each patient and the experience of interventional radiologists.
  Other Names: TACE
  Arms: Sorafenib plus TACE

SUMMARY:
This trial is a multi-center, phase III, randomized (1:1) clinical trial. The aim is to explore the efficacy and safety of Sorafenib combined with transarterial chemoembolization as adjuvant treatment for resectable advanced hepatocellular carcinoma, compared with Sorafenib alone. The primary endpoint is recurrence-free survival. This trial planned to recruit 158 patients who received curative hepatic resection with resectable advanced hepatocellular carcinoma. The patients will be randomized into Sorafenib group and Sorafenib+TACE group as 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Primary hepatocellular carcinoma without any treatments.
2. Received curative hepatic resection
3. ECOG score 0-1
4. Child-Pugh grade A
5. Sufficient liver and kidney function

Exclusion Criteria:

1. Diffused lesions; tumor thrombosis in SMV or IVC.
2. Extra-hepatic metastasis.
3. Contraindication of TACE, like portal-systemic shunt, obvious atherosclerosis, etc.
4. Allergic to the contrast agent of TACE
5. Dysfunction of liver, kidney or bone marrow.
6. Concomitant other malignant tumor or HIV infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2021-09-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 2 years
  Recurrence-free survival indicates the interval between randomization and tumor recurrence or death.[0-2 years] Longer RFS time indicates better prognosis.

SECONDARY OUTCOMES:
Overall survival | 2 years
  Overall survival indicates the interval between randomization and death.[0-2years]Longer OS time indicates better prognosis.
Time to recurrence | 2 years
  Time to recurrence indicates the interval between randomization and tumor recurrence.[0-2years]Longer TTR time indicates better prognosis.
Severe adverse events | 2 years
  Incidence rate of severe adverse events. [0-100%]. lower rate indicates more safety of the treatment
Quality of life | 2 years
  Questionnaire score of EORTC-QOL. Higher score indicates better quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peng Z, Fan W, Liu Z, Xiao H, Wu J, Tang R, Tu J, Qiao L, Huang F, Xie W, Zhuang W, Guo W, Li S, Hua Y, Shen S, He Q, Li D, Li J, Kuang M. Adjuvant Transarterial Chemoembolization With Sorafenib for Portal Vein Tumor Thrombus: A Randomized Clinical Trial. JAMA Surg. 2024 Jun 1;159(6):616-624. doi: 10.1001/jamasurg.2024.0506. PMID 38568599